CLINICAL TRIAL: NCT06712238
Title: Evaluation The Effect of NB-UVB and Methotrexate on The Level of Serum Gelsolin in Psoriatic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Nourhan Salah Mohamed, Resident of Dermatology, Venereology and Andrology, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nourhan Salah
Record Dates: First submitted 2024-11-20; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-06

CONDITIONS: Psoriatic Conditions
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: (Narrow Band Ultraviolet B) (Active Comparator): About 12 patients will expose to 24 sessions of Narrow Band Ultraviolet B (NB-UVB) radiation (initial dose of 130 - 400 mJ / cm2 ) selected according to skin for 3 month.
  Interventions: Procedure: NB-UVB
- Group B: (Methotrexate ) (Active Comparator): About 12 patients will receive Methotrexate tablets (MTX) in dose of (0.3 mg/kg/week) along with folic acid (5 mg/day) for 3 month.
  Interventions: Procedure: NB-UVB
- Group C: (Methotrexate and Narrow Band Ultraviolet B) (Active Comparator): About 12 patients will undergo the treatment by both Methotrexate tablets (MTX) and Narrow Band Ultraviolet B( NB-UVB) radiation.for 3 month.
  Interventions: Procedure: NB-UVB
- Group D (Control Group) (Active Comparator): About 12 patients apparently healthy individuals as control group.and will not take any medication
  Interventions: Procedure: NB-UVB

INTERVENTIONS:
Procedure: NB-UVB — Comparison between serum Level of Gelsolin (GSN) in Psoriatic Patients and controls and correlate its level with PASI.
  Other Names: Methotrexate

SUMMARY:
Psoriasis is a common chronic, immune-mediated, skin disease with a significantly negative impact on patients' quality of life. It is one of papulosquamous diseases defined by erythematous plaques with silvery scales.

The interplay among cytokines released by dendritic, Th1, Th2, and Th17 cells leads to the clinical manifestations seen in psoriasis. Although discovering novel biomarkers for psoriasis is challenging step., it may play an essential role in diagnosis, severity assessment and prediction of treatment outcome and prognosis of the disease

DETAILED DESCRIPTION:
The protein expression of gelsolin- which is an actin scavenger controlling cytoskeletal remodeling, cell morphology, differentiation, movement, and apoptosis- has been found to be significantly decreased in several pathological conditions including neurodegenerative diseases, inflammatory disorders, and cancers.

Gelsolin (GSN) is a member of the GSN protein family, the main function of it is to cut and seal actin filaments to regulate the cytoskeleton and participate in a variety of biological functions.

Low serum gelsolin levels are linked to the severity of psoriasis, suggesting that gelsolin may help in assessing the severity of the disease and how it responds to treatment.

Methotrexate (MTX) is the first-choice drug when phototherapy or retinoid treatment are not effective in psoriatic patients.

It is a cytotoxic drug with powerful anti-proliferative and anti-inflammatory effects that has gained prominence in treating inflammatory diseases one of them is psoriasis.

Narrowband (NB) UVB phototherapy is a common line of treatment in psoriasis. It was proven to be more effective than broadband UVB and safer and/or more practicable than psoralen_UVA in treatment of psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe plaque psoriasis.
* No restriction of age, race nor occupation.

Exclusion Criteria:

* History of psoriasis treatment with systemic and biological agents prior to the study for at least 3 months.
* Pregnancy and lactation.
* Infections.
* Patients with chronic diseases: hepatic disorders, hematologic diseases, chronic renal failure or cancer.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Treatment of the Psoriasis | 3 months
  About 36 patients suffering from Psoriasis and will be treated by exposing to Narrow band ultraviolet B radiation (initial dose of 130 - 400 mJ / cm2 selected according to skin phototype and gradual increase after each session ), and taking Methotrexate tablets in dose of (0.3 mg/kg/week) along with folic acid (5 mg/day) .
Serum Gelsolin Evaluation | 3 Months
  Evaluation the Serum Gelsolin level in Psoriatic Patients after treatment by Narrow band ultraviolet B and taking Methotrexate tablets.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Adam Ali El Taieb, Professor, Study Chair — Dermatology, Venereology and Andrology.Faculty of Medicine, Aswan University
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided